CLINICAL TRIAL: NCT05886179
Title: Factors Associated With COVID-19 in Children Aged 0-15 Years in Niger, 2020
Brief Title: COVID-19 IN CHILDREN IN NIGER, 2020
Status: Completed | Type: Observational
Sponsor: Centre de Recherche Médicale et Sanitaire (Other)
Responsible Party: Principal Investigator, IDE AMADOU Habibatou, Doctor, Centre de Recherche Médicale et Sanitaire
Other Study IDs: CERMES
Record Dates: First submitted 2023-05-31; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: to Contribute to a Better Control of COVID-19 in Children in Niger
Keywords: factors, COVID-19, children, database, Niger
MeSH Terms: conditions — COVID-19 | interventions — Cross-Sectional Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: cross-sectional study — analytical cross-sectional study with retrospective collection of epidemiological surveillance data on COVID-19 in Niger.

SUMMARY:
On January 30, 2020, the WHO declared COVID-19 a global health emergency. Children were affected with less severe forms. Niger had implemented measures in a context where children are a source of contamination. The objective was to determine the factors associated with COVID-19 in children in Niger from February to August 2020 through an analysis of the national database.

DETAILED DESCRIPTION:
We conducted an analytical cross-sectional study including all COVID-19 suspects in the database. We used Excel and Epi Info 7.2.4. software for data extraction and analysis. Frequencies and proportions were calculated, we estimated in a logistic regression the OR of association with their 95% confidence interval, the factors associated with COVID-19 at the threshold of p<0.05.

Results: Of 572 notified suspected COVID-19 cases in children aged 0-15 years, 11.36% were positive. The median age of infected children was 10 years [IQR: 5- 13 years]. The sex ratio of males to females was 2.1. Children aged 11-15 years were 49.2%, 61.5% resided in Niamey, 4.6% had comorbidities. The notion of travel was 12.3% and 40% had a notion of contact, 24.4% had a fever, 23.2% had a cough, 18% were hospitalized and the case fatality was 1.5%. In etiological analysis, the factors associated with COVID-19 were sex ORa= 0.51 [0.28-0.93] p=0.028, the presence of symptoms ORa= 2.29 [1.23-4.25] p=0.008 and the notion of contact ORa= 0.32 [0.13-0.77] p=0.011.

exposed children were sensitive to COVID-19, all age groups were affected with a male predominance. We recommend barrier measures adapted to young people, early detection and management of infected children.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0-15 years suspected of having COVID-19 whose data were in the DSRE database were included

Exclusion Criteria:

* Children whose data is not complete

Ages: 0 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This was an analytical cross-sectional study with retrospective collection of epidemiological surveillance data on COVID-19 in Niger. The study period spanned six (6) months from February 25 to August 28, 2020. Children aged 0-15 years suspected of having COVID-19 whose data were in the DSRE database were included. We used the data extraction form that served as a secondary database containing only our variables of interest.
Sampling Method: Non-Probability Sample
Enrollment: 572 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
data base analysis | May 2021
  The first step concerned the descriptive part where the frequencies, proportions, means and extreme values of the variables were calculated. Some of these variables were presented in the form of tables and graphs.

CONTACTS AND LOCATIONS:
Locations (1):
- IDE AMADOU Habibatou, Niamey, Niger

IPD SHARING:
Plan to Share IPD: No
What is IPD ?